CLINICAL TRIAL: NCT01917851
Title: Evaluate the Accuracy of the NBM200 for Noninvasive Hemoglobin Measurements on Obstetric/Gynecological Patients.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: OrSense, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: NBMHB-PRS-2
Record Dates: First submitted 2013-07-28; First posted 2013-08-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-07

CONDITIONS: Anemia
Keywords: Accurate; Hb; noninvasive measurement
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to define the precision, accuracy and variability of the NBM-200 system in non invasive blood Hemoglobin (Hb) measurements relative to the laboratory blood analyzer by comparing two consecutive Hb values obtained by the NBM system to venous values.

DETAILED DESCRIPTION:
Each subject will be placed in a comfortable position in a temperature regulated room. Participants will have two consecutive non invasive (NBM) measurements taken which involves inserting the thumb into a ring shaped sensor. After each non invasive measurement the sensor will be removed. Each measurement takes approximately 85 seconds and involves the finger cuff inflating (to over systolic pressure) and deflating several times in quick successions in order to measure and calculate the Hb values. The two non invasive measurements will be performed using the same finger. After the NBM system testing is complete and recorded, the subject will have a venous (venipuncture) blood sample collected in order to provide two blood tests performed on two different models of routine automated CBC or Hb blood analyzers.

ELIGIBILITY:
Inclusion Criteria:

* Female volunteers aged 18 years and over.
* Any patient subject to CBC testing according to OBGYN standard care and clinical judgment.

Exclusion Criteria:

* Participants under the age of 18 years
* Significant deformity, degenerative changes or edema of the thumb or index fingers
* Localized infection, ulceration or skin breaks involving the fingers
* Low peripheral body temperature (tissue perfusion) <36.0˚C
* Vascular disease or Raynaud's phenomenon affecting the fingers
* Participants who are unable to give informed written consent

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-04; Primary Completion 2013-08 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Compare the Hb values from the NBM200 series against the Hb from the lab blood analyser on obstetric/gynecological patients. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Eran Hadar, MD, Principal Investigator — Rabin Medical Center